CLINICAL TRIAL: NCT04376502
Title: Phase II Trial of Immune Checkpoint Inhibitor and Novel in Situ Radiation "Booster Shot" Tumor Vaccination in Patients With Metastatic Carcinoma
Brief Title: Immune Checkpoint Inhibitor and MR-guided SBRT for Limited Progressive Metastatic Carcinoma.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: Baptist Health South Florida (Other)
Collaborators: Viewray Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-CHU-001
Record Dates: First submitted 2020-05-01; First posted 2020-05-06 (Actual); Results first posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Carcinoma
Keywords: radiation
MeSH Terms: conditions — Carcinoma | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: Radiation therapy for all subjects will consist of treating one tumor of the treating physician's preference (40 Gray (GY) in 5 fractions), and after a 1-week interval during which Immune checkpoint inhibitor is continued alone, radiation therapy will be given to a second and separate tumor (30 Gy in 5 fractions).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- radiation therapy (RT) (Other): RT for all subjects will consist of treating one tumor of the treating physician's preference (40 Gy in 5 fractions), and after a 1-week interval during which Immune checkpoint inhibitor (ICI) is continued alone, RT will be given to a second and separate tumor (30 Gy in 5 fractions).
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — Radiation therapy for all subjects will consist of treating one tumor of the treating physician's preference (40 Gray (Gy) in 5 fractions), and after a 1-week interval during which ICI is continued alone, radiation therapy will be given to a second and separate tumor (30 Gy in 5 fractions).

SUMMARY:
This is an open label single arm phase 2 clinical trial in patients with metastatic solid malignancy of any histology who have previously experienced limited progression in at least 1 and up to 5 lesions while on immune checkpoint inhibitors monotherapy.

DETAILED DESCRIPTION:
All potential subjects are required to undergo screening evaluation to determine eligibility within 28 days of study enrollment.

Eligible subjects will continue the same immune checkpoint inhibitors on which they experienced limited progression and will also receive radiation therapy. radiation therapy for all subjects will consist of treating one tumor of the treating physician's preference, and after a 1-week interval during which immune checkpoint inhibitor is continued alone, radiation therapy will be given to a second and separate tumor. No additional radiation therapy will be delivered. immune checkpoint inhibitors will be continued until disease progression or unacceptable toxicity. Diagnostic imaging studies will be performed to determine treatment response at baseline/screening, 8 weeks after initiation of radiation therapy to the first lesion and every 8 weeks thereafter.

Peripheral blood mononuclear cell composition will be evaluated at various time points within 14 days of starting radiation therapy, on Day 8 (1 week after starting radiation therapy to the first lesion), Day 23 (1 week after starting radiation therapy to the second lesion), and 8 weeks after treatment initiation.

A total of 52 subjects will be enrolled on this trial. The expected rate of accrual is 2 patients per month at a single institution over 26 months.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age at the time of study entry.
2. Eastern Cooperative Oncology Group performance status of 0, 1, or 2.
3. Life expectancy of .12 weeks as estimated by the treating physician.
4. Metastatic carcinoma confirmed by biopsy or imaging study if biopsy is not deemed feasible.
5. Most recent anti-cancer therapy consists of a single ICI drug including but not limited to ipilimumab, nivolumab, pembrolizumab, atezolizumab.
6. Radiographic evidence of progression while on a single ICI drug in 1 and up to 5 lesions.
7. Eligible to continue ICI during and after radiation therapy.
8. 3 radiographically distinct and measurable lesions (primary and/or metastatic lesions) by RECIST 1.1 criteria, with .3 lesions separated from each other by .5 cm
9. Subjects must consent to all study procedures described in the protocol including radiographic evaluation and blood draws.
10. Immunosuppressive doses of systemic medication including steroids must be discontinued at least 14 days prior to the start of radiation therapy.
11. Adequate normal organ and marrow function
12. Female subjects must either be of non-reproductive potential (i.e., post-menopausal by history: .60 years old and no menses for .1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy), have a negative serum pregnancy test within 14 days of study enrollment, and not be breastfeeding.

Exclusion Criteria:

1. Any contraindication to having an MRI scan.
2. Chemotherapy, biologic agent, investigational therapy, or radiation therapy given within 14 days of study enrollment.
3. Symptomatic or uncontrolled brain metastasis requiring treatment.
4. The need for palliative radiation therapy to a non-target lesion prior to radiation therapy to one of 2 target lesion on this study.
5. Prior radiation therapy to any lesion that would receive radiation therapy on this protocol.
6. Prior radiation therapy to a lesion located within 4 cm of previously irradiated structures: spinal cord that previously received >45 Gy; brachial plexus that previously received >45 Gy; small/large intestine or stomach that previously received >45 Gy; prior total lung V20 >30%.
7. Prior radiation therapy that could lead to an unacceptably high risk of clinically significant normal tissue injury due to high cumulative normal tissue dose as determined by the investigator.
8. History of any primary malignancy with the exception of

   1. Malignancy treated with curative intent and with no known active disease for at least 3 years before enrollment on this study.
   2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
   3. Adequately treated carcinoma in situ without evidence of disease (i.e. cervical carcinoma in situ; superficial bladder cancer).
9. Any unresolved toxicity (Common Terminology Criteria for Adverse Events version 5.0 > grade 2) from previous anti-cancer therapy. Subjects with irreversible toxicity that is not reasonably expected to worsen by treatment on this study are permitted to enroll on this study.
10. Active or prior documented autoimmune disease within the past 2 years. Subjects with vitiligo, type I diabetes mellitus, Graves disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
11. Subjects requiring systemic corticosteroid (>10 mg daily prednisone equivalent) or other immunosuppressive medication within 14 days of study enrollment.
12. Contraindication to IV contrast despite premedication for iodine allergy, which would limit the ability to assess radiographic response to study treatment.
13. Prior allogeneic organ transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-04-08 (Actual); Primary Completion 2023-06-16 (Actual); Study Completion 2023-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Chuong, MD, Principal Investigator — Miami Cancer Institute (MCI) at Baptist Health, Inc.
Locations (1):
- Miami Cancer Institute at Baptist Health South Florida, Miami, Florida, United States

REFERENCES:
- See also: Miami Cancer Institute website — https://baptisthealth.net/cancer-care/home

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Radiation Therapy (RT)
Started | 12
Completed | 11
Not Completed | 1
Not completed — Deemed ineligible after being enrolled | 1

BASELINE CHARACTERISTICS:
Arm/Group | Radiation Therapy (RT)
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.92 (9.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Overall Response Rate (ORR) According to RECIST 1.1 Criteria
Description: ORR is defined as the percent of participants who have a partial response (PR) or complete response (CR) to therapy of non-irradiated lesions according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria assessed on CT imaging. CR is defined as the disappearance of all target and non-target lesions. PR is defined as at least a 30% decrease from baseline in the sum of the longest diameters of target lesions AND for non-target lesions, no progression of existing lesions or appearance of new lesions.
Time Frame: 6 months
Population: Six participants did not receive 6-month imaging and response evaluation. Five were taken off study due to disease progression (two), new AE that made them ineligible to continue (one), other ineligibility (one), or expiration (one). One participant had missed imaging.
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy (RT)
Number analyzed (Participants) | 6
Participants | 1

2. Secondary Outcome: Number of Treatment Related Adverse Events
Description: Treatment related adverse events are defined as those possibly, probably, or definitely related to the study treatment. These events will be tabulated and reported by grade of severity.
Time Frame: through study completion, an average of 1 year
Population: One participant was deemed ineligible after being considered enrolled and was thus withdrawn.
Measure: Number; unit: events
Arm/Group | Radiation Therapy (RT)
Number analyzed (Participants) | 11
events
  Mild (Grade 1) | 19
  Moderate (Grade 2) | 7
  Severe (Grade 3) | 6
  Life-threatening (Grade 4) | 0
  Death (Grade 5) | 0

3. Secondary Outcome: Change in Immune-related ORR (irORR) According to Immune-related Response Criteria (irRC)
Description: irORR is the percent of patients with best overall response of irCR or irPR from the start of the study until 6 months later. Only index and measurable new lesions are taken into account in irRC and response is defined over at least 4 weeks. irCR is defined as the disappearance of all lesions in two observations at least 4 weeks apart. irPR is defined as at least 50% decrease in tumor burden compared with baseline in two observations at least 4 weeks apart.
Time Frame: 6 month
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy (RT)
Number analyzed (Participants) | 6
Participants | 1

4. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time from when CR or PR is first determined until the first date of documented progressive disease (PD) or death, whichever occurs first.
Time Frame: 6 month
Population: Only two participants ever had PR. None had CR. Out of the two participants with PR, one did not have progression during the time points when response was assessed, thus was not included in this calculation.
Measure: Number; unit: days
Arm/Group | Radiation Therapy (RT)
Number analyzed (Participants) | 1
days | 55

5. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the percent of participants who are alive at the end of the study. Death due to any cause will be considered.
Time Frame: 2 years
Population: One participant was deemed ineligible after being considered enrolled and was thus withdrawn.
Measure: Count of Participants; unit: Participants
Arm/Group | Radiation Therapy (RT)
Number analyzed (Participants) | 11
Participants | 5

6. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the amount of time from first treatment to disease progression or death from any cause.
Time Frame: 6 month
Population: One participant was deemed ineligible after being considered enrolled and was thus withdrawn.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Radiation Therapy (RT)
Number analyzed (Participants) | 11
months | 2.5 [1.0 to NA] — Upper bound was not reached for time to event analysis due to lack of enough events observed in the study population by the end of follow-up. Specifically, due to small sample size to start, compounded by censoring of data, many patients did not have the event. Therefore, the upper bound of the 95% confidence interval could not be calculated.

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Radiation Therapy (RT)
All-Cause Mortality (participants affected / at risk) | 6/11
Serious Adverse Events (participants affected / at risk) | 3/11
Other Adverse Events (participants affected / at risk) | 9/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Therapy (RT) (N=11)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Hypotension (Vascular disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiation Therapy (RT) (N=11)
Fatigue (General disorders) | 5 (10)
Nausea (Gastrointestinal disorders) | 4 (5)
Infections and infestations - Other, COVID-19 (Infections and infestations) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Abdominal Pain (Gastrointestinal disorders) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (4)
Edema limbs (General disorders) | 2 (2)
Lung infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Peripheral neuropathy (Nervous system disorders) | 2 (2)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Weight loss (Investigations) | 2 (2)
Aspartate aminotransferase increase (Investigations) | 1 (4)
Alanine aminotransferase increase (Investigations) | 1 (3)
Dermatitis radiation (Injury, poisoning and procedural complications) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (2)
Ascites (Gastrointestinal disorders) | 1 (1)
Bacteremia (Infections and infestations) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Generalized edema (General disorders) | 1 (1)
Generalized muscle weakness (General disorders) | 1 (1)
Hepatobiliary disorders - Other, Biliary ductal dilation (Hepatobiliary disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Infections and infestations - Other, Metapneumovirus (Infections and infestations) | 1 (1)
Investigations - Other, Hyperbilirubinemia (Investigations) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Tremor (Nervous system disorders) | 1 (1)
Watering eyes (Eye disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated early because of poor enrollment. Because the study did not accrue the intended sample of participants, there was not enough power to conduct statistical analysis or calculate accurate estimates.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-22): https://cdn.clinicaltrials.gov/large-docs/02/NCT04376502/Prot_SAP_000.pdf